CLINICAL TRIAL: NCT02092363
Title: A Phase 1b Dose Escalation Study of OMP-54F28 in Combination With Paclitaxel and Carboplatin in Patients With Recurrent Platinum-Sensitive Ovarian Cancer
Brief Title: Dose Escalation Study of OMP-54F28 in Combination With Paclitaxel and Carboplatin in Patients With Recurrent Platinum-Sensitive Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54F28-003
Record Dates: First submitted 2014-02-19; First posted 2014-03-20 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Ovarian Cancer
Keywords: Platinum-Sensitive Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — OMP-54F28; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: OMP-54F28, Paclitaxel and Carboplatin (Experimental)
  Interventions: Drug: OMP-54F28, Paclitaxel and Carboplatin

INTERVENTIONS:
Drug: OMP-54F28, Paclitaxel and Carboplatin
  Other Names: OMP-54F28; Paclitaxel; Carboplatin

SUMMARY:
This is an open-label Phase 1b dose-escalation study to assess the safety, tolerability, and PK of OMP-54F28 when combined with paclitaxel and carboplatin. OMP-54F28 will be administered IV on Days 1 of each 21-day cycle. Paclitaxel (175 mg/m2) and carboplatin (AUC = 5 mg/mL • min) will be administered IV on Day 1 of each cycle. A total of 6 cycles of paclitaxel and carboplatin will be given. Additional cycles may be given as per institutional standard of care after discussion with the Medical Monitor. Treatment with OMP-54F28 will continue after completion of treatment with paclitaxel and carboplatin. The planned dose levels of OMP-54F28 are 5 and 10 mg/kg.

DETAILED DESCRIPTION:
Depending on safety in this study, additional lower or intermediate dose levels may be evaluated. Depending on emerging safety data from the Phase 1a study 54F28-001 with continuing dose escalation, additional higher dose levels of OMP-54F28 may be evaluated in this study. Alternative dosing schedules of OMP-54F28 may be explored based on emerging nonclinical and clinical data for safety, PD, PK and efficacy. The starting dose for a new dosing schedule will be chosen to result in an AUC equivalent to the highest dose level that cleared on the previously studied dosing schedule. No dose escalation of OMP-54F28 will be allowed within a dose cohort.

Once the maximum tolerated dose (MTD) or maximum administered dose (MAD) has been determined, up to 10 patients may be enrolled in the cohort-expansion phase to better characterize the safety, tolerability and PK of OMP-54F28 combined with paclitaxel and carboplatin. Up to approximately 34 patients may be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥18 years
* Histologically documented ovarian, primary peritoneal or fallopian tube cancer
* Recurrent platinum-sensitive disease, defined as disease progression ≥6 months after completing a minimum of 4 cycles of a platinum-containing regimen
* Availability of FFPE tumor tissue, either archival or obtained at study entry through fresh biopsy

  o Tumor tissue from fine needle aspiration is not acceptable.
* ECOG performance status of 0 or 1
* All acute treatment-related toxicity from prior therapy must have resolved to Grade ≤ 1 prior to study entry
* Adequate hematologic and end-organ function
* Evaluable or measurable disease per RECIST v1.1
* For women of childbearing potential, agreement to use two effective forms of contraception

Exclusion Criteria:

* Non-epithelial ovarian carcinoma, including malignant mixed Mullerian tumors
* Prior treatment with paclitaxel and carboplatin for recurrent platinum-sensitive ovarian cancer
* Treatment with any anti-cancer therapy, including radiotherapy, chemotherapy, biologic therapy, or herbal therapy within 3 weeks or 5 half-lives (for systemic agents), whichever is shorter
* Known hypersensitivity to any component of study treatments that resulted in drug discontinuation
* Grade ≥ 2 sensory neuropathy
* Uncontrolled seizure disorder or active neurologic disease
* Untreated brain metastases
* Leptomeningeal disease as a manifestation of cancer
* Active infection requiring antibiotics
* Bisphosphonate therapy for symptomatic hypercalcemia
* Known history of clinically significant liver disease, including active viral hepatitis and cirrhosis
* Significant intercurrent illness including, but not limited to, unstable angina pectoris, and cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements
* Pregnancy, lactation, or breastfeeding
* Known HIV infection
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Concurrent use of therapeutic warfarin
* New York Heart Association Classification III or IV
* Known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the first dose of study treatment or anticipation of need for major surgical procedure during the course of the study
* Osteoporosis based on a T-score of <-2.5 at the left or right total hip, left or right femoral neck or lumbar spine (L1-L4) as determined by DEXA scan
* Bone metastases and one of the following:

  * Prior history of a pathologic fracture
  * Lytic lesion requiring an impending orthopedic intervention
  * Lack of treatment with a bisphosphonate or denosumab
* Treatment with a thiazolidinedione PPAR gamma inhibitor; e.g. Actos® (pioglitazone) and Avandia® (rosiglitzone)
* Active treatment with an oral or IV glucocortocoid for ≥4 weeks at a daily dose equivalent to or greater than 7.5 mg of oral prednisone
* Fasting β-CTX of >1000 pg/mL
* Metabolic bone disease, such as hyperparathyroidism, Paget's disease or osteomalacia

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-01; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of OMP-54F28 in combination with paclitaxel and carboplatin in patients with recurrent platinum-sensitive ovarian cancer | Subjects will be treated and observed for DLT through the end of the first cycle (from Day 0 - 21)
  The maximum tolerated dose (MTD) will be determined in patients treated with OMP-54F28/paclitaxel/carboplatin (from Day 0 - 21)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - OU Medical Center Laboratory, Oklahoma City, Oklahoma
  - The University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Fox-Chase Cancer Center, Philadelphia, Pennsylvania